CLINICAL TRIAL: NCT05023226
Title: Effectiveness of Recruitment Maneuvers and Lung Protective Ventilation Strategy in ARDS
Acronym: ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AUH-CT-ZK01
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: ARDS
Keywords: Acute respiratory distress syndrome (ARDS); Recruitment maneuvers (RM); Oxygenation index(OI); Lung ultrasound score(LUS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPVS group (Placebo Comparator): The general ventilator setting.
  Interventions: Procedure: LPVS
- LPVS + RM group (Experimental): Recruitment maneuver.
  Interventions: Procedure: RM; Procedure: LPVS

INTERVENTIONS:
Procedure: RM — RM refers to that under FiO2=100% oxygen concentration and fixed inspiratory pressure (15cmH2O), the PEEP starts from 10 cmH2O and increases at a pressure of 5 cmH2O every minute until the Peak inspiratory Pressure(PIP) reaches 55cmH2O, and the level was fixed to 40 seconds in each increment. Then, the ventilator was transferred to PEEP-titration phase, the PEEP was adjusted to 25 cm H2O, and it was reduced by increments of 5 cm H2O each time. The each increment was fixed to 5 minutes till the end-maneuver PEEP.
  Other Names: Recruitment maneuver
  Arms: LPVS + RM group
Procedure: LPVS — LPVS was used by the pressure-controlled mode and the PEEP was titrated by the level of FiO2 to keep the saturation of oxygen (SaO2) more than 90%. The level of pressure control was adjusted to maintain low tidal volume (6-8 mL/kg predicted body weight [PBW]) strategy. The respiratory rate and tidal volume were setting to avoid unstable hemodynamic data and adjusted by blood gas data and lung mechanics.
  Other Names: Lung protective ventilation strategies

SUMMARY:
The study was designed to comparison the effectiveness of recruitment maneuvers(RM) and lung protective ventilation strategy(LPVS) for patients with moderate to severe ARDS.

ARDS patients were randomly divided into two groups, the experimental group (LPVS+RM group) and the control group (LPVS group). The method of RM refers to that under FiO2=100% oxygen concentration and fixed inspiratory pressure (15cmH2O), the PEEP starts from 10 cmH2O and increases at a pressure of 5 cmH2O every minute until the Peak inspiratory Pressure(PIP) reaches 55cmH2O, and the arterial blood oxygen is monitored at the same time. The pressure point when the partial pressure of arterial oxygen PaO2+PaCO2≧400mmHg is the best PEEP. The primary endpoint indicators were oxygenation index(OI) and lung ultrasound score(LUS) from day 1 to day 7. The secondary outcome indicators were the ventilator days, length of stay in the ICU (days), and ICU mortality.

DETAILED DESCRIPTION:
ARDS patients were randomly divided into two groups, the experimental group (LPVS+RM group) and the control group (LPVS group). The method of RM refers to that under FiO2=100% oxygen concentration and fixed inspiratory pressure (15cmH2O), the PEEP starts from 10 cmH2O and increases at a pressure of 5 cmH2O every minute until the Peak inspiratory Pressure(PIP) reaches 55cmH2O, and the arterial blood oxygen is monitored at the same time. The pressure point when the partial pressure of arterial oxygen PaO2+PaCO2≧400mmHg is the best PEEP. The primary endpoint indicators were oxygenation index(OI) and lung ultrasound score(LUS) from day 1 to day 7. The secondary outcome indicators were the ventilator days, length of stay in the ICU (days), and ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 70 years old.
* Patients with hypoxemia receiving endotracheal mechanical ventilation therapy.
* The ARDS diagnostic criteria of Berlin Definition, arterial oxygen tension [PaO2]/fractional inspired oxygen [FiO2] ratio (PaO2/FiO2) <200 mm Hg, recent appearance of bilateral pulmonary infiltrates consistent with edema and no clinical evidence of left atrial hypertension.
* Within 72 hours after ARDS diagnosis.

Exclusion Criteria:

* Pregnancy.
* Participate in other interventional trials at the same time during the acceptance period.
* Severe trauma combined with rib fracture or pneumothorax, subcutaneous emphysema, and mediastinal air accumulation within three months.
* Severe chronic respiratory diseases that require long-term use of oxygen therapy or home mechanical ventilation.
* Have a history of cachexia or terminal cancer.
* Use immunosuppressants, chemotherapy or radiation therapy.
* Contraindications for hypercapnia, such as patients with acute brain injury due to intracranial hypertension or craniotomy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index(OI) | Baseline - 72 hrs after enrollment
  Difference in OI between baseline and 72 hrs after enrollment 【The oxygenation index assesses the intensity of ventilatory support that is needed to maintain adequate oxygenation. The formula is: Oxygenation index = (FiO2 x PAW) / PaO2. The lower the OI(<25) the better the outcome】
Lung ultrasound score(LUS) | Baseline - 72 hrs after enrollment
  Difference in LUS between baseline and 72 hrs after enrollment 【LUS is a score that measures lung aeration, score ranging from 0 to 36 points, the higher the score is mean the worse the ventilation of the lungs】

SECONDARY OUTCOMES:
Ventilator days | Removal of endotracheal tube day - Insertion endotracheal tube day + 1 day
  Removal of endotracheal tube without ventilator support days
Length of stay in the ICU (days) | Transfer out of ICU day - Admission to ICU day + 1 day
  Total days of admission ICU
ICU mortality | During ICU course
  In ICU death after admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Zi-Tin Kuan, RN, Study Director — Asia University Hospital
Locations (1):
- Asia University, Taichung, Wufeng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chung FT, Lee CS, Lin SM, Kuo CH, Wang TY, Fang YF, Hsieh MH, Chen HC, Lin HC. Alveolar recruitment maneuver attenuates extravascular lung water in acute respiratory distress syndrome. Medicine (Baltimore). 2017 Jul;96(30):e7627. doi: 10.1097/MD.0000000000007627. PMID 28746224
- See also: doi: 10.1097/MD.0000000000007627 — https://doi.org/10.1097/MD.0000000000007627